CLINICAL TRIAL: NCT03879902
Title: The Characteristics of Falls in Community-dwelling Older Adults in Hong Kong and Its Potential Predictors
Brief Title: The Characteristics of Falls and Its Potential Predictors
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Timothy Kwok, Professor, Chinese University of Hong Kong
Other Study IDs: 2018.076
Record Dates: First submitted 2019-02-24; First posted 2019-03-19 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Fall Patients
Keywords: fall; elderly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective study to examine the fall characteristics among elderly faller in Hong Kong and the potential predictors of falls incidence.

DETAILED DESCRIPTION:
This will be a prospective study. One thousand and five hundred older fallers would be recruited. Baseline assessments would be conducted to examine potential fall risk factors and the fall history. The subjects would be followed up for 1 year for fall incidence. This study conforms to the ethical principles of the World Medical Association Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 or older
* able to ambulate with a Functional Ambulation Category (FAC) score ≥ 3
* able to walk for ≥ 10 meters
* history of falls in the past 12 months
* living in the community
* able to understand Chinese

Exclusion Criteria:

* blindness

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community-dwelling older adults with fall history
Sampling Method: Non-Probability Sample
Enrollment: 2101 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Number of falls | 1 year
  Prospective fall data will be collected through telephone follow-up for 1 year. The number of fall during the follow-up period and the circumstances while the falls occur would be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Kwok, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong Jockey Club Centre of Osteoporosis Care and Control, Hong Kong, Hong Kong